CLINICAL TRIAL: NCT01494597
Title: Effect of Multiple Doses of Isavuconazole on the Pharmacokinetics of a Single Dose of Cyclosporine: A Phase 1, Open-Label, Sequential Study in Healthy Adult Subjects
Brief Title: Drug Interaction Study of Isavuconazole and Cyclosporine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Collaborators: Basilea Pharmaceutica International Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 9766-CL-0022
Record Dates: First submitted 2011-12-15; First posted 2011-12-19 (Estimated); Last update posted 2011-12-19 (Estimated); Status verified 2011-12

CONDITIONS: Healthy
Keywords: Isavuconazole; Cyclosporine; Healthy Volunteers; BAL8557; Pharmacokinetics of isavuconazole; Pharmacokinetics of cyclosporine
MeSH Terms: interventions — isavuconazole; Cyclosporine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Isavuconazole and cyclosporine (Experimental): Isavuconazole three times per day (TID) for two days followed by once a day (QD) for 6 days. Cyclosporine single doses on Days 1 and 15.
  Interventions: Drug: isavuconazole; Drug: cyclosporine

INTERVENTIONS:
Drug: isavuconazole — oral
  Other Names: BAL8557
Drug: cyclosporine — oral
  Other Names: Neoral

SUMMARY:
The purpose of this study is to assess the effect of multiple doses of isavuconazole on the pharmacokinetics of cyclosporine in healthy adult subjects.

DETAILED DESCRIPTION:
Subjects will be enrolled to receive a single dose of cyclosporine on Day 1 followed by a 10-day wash-out period (time from cyclosporine dosing to isavuconazole dosing). On Days 11 and 12, isavuconazole will be dosed three times daily (TID). On Days 13 through 18, isavuconazole will be administered once daily (QD). All subjects will be administered a single dose of cyclosporine on Day 15. Subjects will be confined in the study center from Day -1 until Day 5 and from Day 10 until Day 19.

A follow up visit will be scheduled approximately 7 ± 2 days after final dosing of isavuconazole.

Blood and urine samples will be taken at various times during the study.

ELIGIBILITY:
Inclusion Criteria:

* The subject must weigh at least 45 kg and have a body mass index (BMI) of 18 to 32 kg/m2, inclusive
* The subject has a normal 12-lead electrocardiogram (ECG)
* The subject's clinical laboratory test results are within normal limits
* Results for aspartate aminotransferase (AST), alanine aminotransferase (ALT) and total bilirubin must be within the normal range
* If female, the subject agrees to sexual abstinence, or is surgically sterile, postmenopausal (defined as at least 2 years without menses), or using a medically acceptable double barrier method (eg, spermicide and diaphragm, spermicide and condom) to prevent pregnancy and agrees to continue using this method from Screening until three weeks after the follow up visit at the end of study; and is not lactating or pregnant as documented by negative serum pregnancy tests
* If male, the subject agrees to sexual abstinence, is surgically sterile, or is using a medically acceptable method to prevent pregnancy during the study period and for three weeks after the follow up visit at the end of the study

Exclusion Criteria:

* Any clinically significant (as judged by the Investigator) disease history of the following systems: pulmonary, gastrointestinal, cardio-vascular (including a history of clinically significant arrhythmia or clinically significant conduction delays on ECG), hepatic, neuro-logical, psychiatric, renal, genitourinary, endocrine, metabolic, dermatologic, immunologic, hematologic, or malignancy excluding non melanoma skin cancer
* The subject has a history of, or has active psoriasis
* The subject has a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmia or torsade de pointes, structural heart disease, or family history of Long QT syndrome (suggested by sudden death of a close relative at a young age due to possible or probable cardiac causes)
* History of tuberculosis or exposure to anyone known or suspected to have tuberculosis or any illness that might confound the results of the study or pose additional risk in administering study drug to the subject
* The subject has/had a symptomatic, viral, bacterial (including upper respiratory infection), or fungal (non-cutaneous) infection within 1 week prior to clinic admission
* The subject has received a vaccination within the last 30 days prior to study drug administration or plans to receive any vaccinations within 2 weeks after the last dose of study drug
* The subject has a positive result for hepatitis B surface antigen, hepatitis C antibodies, or QuantiFERON®-TB Gold test(s) or is known to be positive for human immunodeficiency virus
* The subject has a known or suspected allergy to any of the components of the trial products or the azole class of compounds or a history of multiple and/or severe allergies to drugs or foods or a history of severe anaphylactic reactions
* The subject is a smoker (any use of tobacco or nicotine containing products) in the last 6 months
* The subject has had treatment with prescription drugs or complementary and alternative medicines within 14 days prior to study drug administration, or over-the-counter medication within 1 week prior to Day -1, with the exception of acetaminophen up to 2 g/day
* The subject has received an experimental agent within 30 days or 5 half-lives, whichever is longer, prior to Day -1
* The subject has had any significant blood loss, donated one unit (450 mL) of blood or more, or received a transfusion of any blood or blood products within 60 days or donated plasma within 7 days prior to clinic admission
* The subject has taken part in strenuous exercise within 3 days before dosing in this trial
* The subject anticipates an inability to abstain from caffeine or alcohol use for 48 hours prior to clinic admission and throughout the duration of the study; or from grapefruit, grapefruit juice, star fruit, or Seville oranges or any products containing these items from 72 hours prior to clinic admission and throughout the duration of the study
* The subject has a recent history (within the last 2 years) of drug or alcohol abuse, or a positive drug screen
* The subject has any other condition which precludes the subject's participation in the trial

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Composite of Pharmacokinetic (PK) variables for cyclosporine (in whole blood): Area under the concentration-time curve (AUC) from time 0 extrapolated to infinity (AUCinf), AUC from time of dosing to the last quantifiable concentration (AUClast), Cmax | Days 1 and 15

SECONDARY OUTCOMES:
Composite of PK variables for cyclosporine (in whole blood): time to attain Cmax(tmax), apparent volume of distribution (Vz/F), apparent body clearance after oral dosing (CL/F), and apparent terminal elimination half-life (t 1/2) | Days 1 and 15
PK variable for Isavuconazole (in plasma): trough concentration (Ctrough) | Day 13 and Days 17 through 19
Composite of PK variables for Isavuconazole (in plasma): AUC during time interval between consecutive dosing (AUCtau), maximum concentration (Cmax),and time to attain Cmax (tmax) | Days 14 and 15

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Global Development
Locations (1):
- Covance, Madison, Wisconsin, United States